CLINICAL TRIAL: NCT00482235
Title: A Study of MK0359 in Patients With Chronic Obstructive Pulmonary Disease (COPD)(0359-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0359-016; 2007_569
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: MK0359

SUMMARY:
A study to test the effect of MK0359 in lessening the symptoms of COPD as compared to salmeterol and placebo.

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 40 and 75
* You have had a history for at least a year of COPD symptoms
* You have a history of smoking one pack of cigarettes per day for 10 years

Exclusion Criteria:

* You have been in a research study with an investigational drug or vaccine in the last 4 weeks.
* You have donated blood in the last 4 weeks.
* You have been hospitalized or had major surgery in the last 4 weeks
* You have been treated in the emergency room within the last 2 months or hospitalized within the last 3 months for your COPD symptoms
* You have a history of heart problems in the last 6 months
* You have a history of stomach problems
* You are unwilling to avoid grapefruit juice throughout the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-12; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lu S, Liu N, Dass SB, Reiss TF, Knorr BA. Randomized, placebo-controlled study of a selective PDE4 inhibitor in the treatment of asthma. Respir Med. 2009 Mar;103(3):342-7. doi: 10.1016/j.rmed.2008.10.024. Epub 2009 Jan 8. PMID 19135348